CLINICAL TRIAL: NCT03305536
Title: Decalcification of the Aortic Valve by Vitamin K2 (Menaquinone-7)
Acronym: DECAV-K2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital St. Georges, Ajaltoun (Other)
Collaborators: Omicron Pharmaceuticals (Industry); Nattopharma ASA (Industry)
Responsible Party: Principal Investigator, Rodolph Frangi, Head of Department of Thoracic and Cardiovascular surgery, Hopital St. Georges, Ajaltoun
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC27082017
Record Dates: First submitted 2017-08-30; First posted 2017-10-10 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Aortic Valve Disease
Keywords: AVD
MeSH Terms: conditions — Aortic Valve Disease | interventions — Vitamin K 2; menaquinone 7; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Active Comparator): 1000 mcg/day of Vitamin K2 + 5000 IU/day Vitamin D3 as a treatment to decalcifiy the valve
  Interventions: Dietary Supplement: Vitamin K2 (Menaquinone 7) + Vitamin D3
- interventional (Active Comparator): 5000 IU/day of Vitamin D3 will be given to measure the progression of the disease along the time of the study
  Interventions: Dietary Supplement: Vitamin K2 (Menaquinone 7) + Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin K2 (Menaquinone 7) + Vitamin D3 — Vitamin K2 + Vitamin D3 arm will be compared with Vitamin D3 arm to slow of reverse the progression of the disease
  Other Names: K2/D3

SUMMARY:
Aortic Stenosis is a common but fatal disease when it becomes symptomatic, specially if not treated. Until now surgery remains the only reliable and effective treatment.

In this study, the investigators will examine the effect of high dose of Menaquinone-7 (MK-7) supplementation (1000 mcg)/day on the progression of the aortic valve disease. The investigators hypothesize that MK-7 supplementation may slow or even reverse the progression of the disease process.

DETAILED DESCRIPTION:
The study is a randomized clinical trial that will use Cardiac Echography and multi-detector computed tomography to compare the changes in the Aortic Valve Calcification Score (AVCS) over 3 years when using:

1. 1000 mcg/d Vitamin K2 (menaquinone-7) + 5000 IU/d Vitamin D3
2. 5000 IU/d Vitamin D3 as a control group

ELIGIBILITY:
Inclusion Criteria:

* AVCS > 300 without aortic valve stenosis requiring operation
* Focus on patients with:

  1. Bicuspid aortic valve
  2. Dialysis or CKD
  3. Statin treatment

Exclusion Criteria:

* Use of Vitamin K antagonist
* Malabsorption Problem
* LVEF < 40%
* A life expectancy < 3 years

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evolution of the Aortic Valve Hemodynamic measured by echography: Change in Gradients in (mm Hg) | 3 years
Evolution of the Aortic Valve Hemodynamic measured by echography: Change in Surface area in (cm2/m2) | 3 years
Evolution of the Aortic Valve Hemodynamic measured by echography: Change in V max in (m/sec) | 3 years

SECONDARY OUTCOMES:
Activation of the MGP measured by the dp-uc MGP level which is a marker of vascular calcification. | 3 years
  1. Lowering of dephosphorelated-undercarboxylated matrix Gla protein (dp-ucMGP picomol/l)
  2. Reduction of the Aortic Valve Calcification Score(AVCS)
  3. Improvement of dyspnea according to the New York Heart Association Classification(NYHA)
  4. Improvement of the quality of life of the patients( physical activity, mobility)
Reduction of the Aortic Valve calcification measured by CT Scan | 3 years
  Reduction of the Aortic Valve Calcification Score (AVCS)
Improvement of dyspnea (at rest and effort) | 3 years
  Improvement of dyspnea according to the New York Heart Association Classification(NYHA)
Improvement of the quality of life of the patients | 3 years
  Every patient have to feel the WHOQOL-BREF, Questionnaire, June 1997, Updated 1/10/2014

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint-George Ajaltoun, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided